CLINICAL TRIAL: NCT02619682
Title: Alternating the Administration of Ixazomib and Lenalidomide as Maintenance Therapy After Autologous Transplant for Treating Multiple Myeloma
Brief Title: Alternating Ixazomib Citrate and Lenalidomide as Maintenance Therapy After Stem Cell Transplant in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Principal Investigator, Leona Holmberg, Professor, Clinical Research Division, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9266; NCI-2015-01861 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); X16064; 9266 (Other: Fred Hutch/University of Washington Cancer Consortium); RG9215039 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2015-11-30; First posted 2015-12-02 (Estimated); Results first posted 2022-07-05 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Plasma Cell Myeloma; Transplant-Related Carcinoma
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ixazomib citrate and lenalidomide) (Experimental): Within 30-120 days after finishing autologous transplant, patients receive ixazomib citrate PO on days 1, 8 and 15. Treatment repeats every 28 days for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients then receive lenalidomide PO QD on days 1-28. Treatment repeats for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients will continue to alternate between ixazomib citrate and lenalidomide every 2 courses for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ixazomib Citrate; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide

INTERVENTIONS:
Drug: Ixazomib Citrate — Given PO
  Other Names: MLN-9708; MLN9708; Ninlaro
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid

SUMMARY:
This phase II trial studies the safety of alternating ixazomib citrate and lenalidomide as treatment to help keep cancer from coming back after stem cell transplant (maintenance therapy) in treating patients with multiple myeloma. Ixazomib citrate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Lenalidomide may stimulate the immune system to attack cancer cells. Giving ixazomib citrate and lenalidomide as maintenance therapy after transplant may prolong the length of time until the cancer returns.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the toxicity of the use of ixazomib (ixazomib citrate) and lenalidomide as maintenance therapy after autologous transplant.

SECONDARY OBJECTIVES:

I. Evaluate the ability to deliver the planned therapy.

II. Assess initial response to therapy.

III. Evaluate the median time to disease progression.

IV. Assess overall survival.

OUTLINE:

Within 30-120 days after completion of autologous transplant, patients receive ixazomib citrate orally (PO) on days 1, 8 and 15 every 28 days for 2 courses, followed by lenalidomide PO once daily (QD) on days 1-28 for 2 courses. Treatment repeats, alternating after every 2 courses, for up to 24 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status and/or other performance status 0, 1, or 2
* Any autologous patient who underwent high dose melphalan (>= 140 mg/m^2) therapy/peripheral blood stem cell (PBSC) rescue for any stage of multiple myeloma and did not participate in another clinical transplant trial whose primary endpoint is also evaluating long-term, disease-free survival or survival; consenting for study between 30 days to 120 days after transplant; earliest can start therapy is 30 days post transplant after recovered from acute toxicity of autologous stem cell transplant (ASCT)
* Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care
* Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject; (periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
* Male patients, even if surgically sterilized (i.e., status post-vasectomy), must agree to one of the following:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject; (periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
* Absolute neutrophil count (ANC) >= 1,000/mm^3
* Platelet count (transfusion independent) >= 75,000/mm^3
* Total bilirubin =< 1.5 x the upper limit of the normal range (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN
* Calculated creatinine clearance >= 30 mL/min

Exclusion Criteria:

* Female patients who are lactating or have a positive serum pregnancy test during the screening period
* Failure to have fully recovered (i.e., =< grade 1 toxicity) from the reversible effects of prior ASCT chemotherapy
* Major surgery within 14 days before enrollment
* Radiotherapy within 14 days before enrollment; if the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of the ixazomib
* History of central nervous system multiple myeloma involvement
* Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months
* Systemic treatment, within 14 days before the first dose of ixazomib, with strong inhibitors of cytochrome P450, family 1, subfamily A, polypeptide 2 gene (CYP1A2) (fluvoxamine, enoxacin, ciprofloxacin), strong inhibitors of cytochrome P450, family 3, subfamily A gene locus (CYP3A) (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort
* Ongoing or active systemic infection, active hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent; patient cannot be allergic to boron
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease; patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection
* Patient has >= grade 2 peripheral neuropathy, or grade 1 with pain on clinical examination during the screening period
* Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial
* Patients with history prior to transplant of progression on lenalidomide therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-12-30 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2025-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leona Holmberg, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: all patients enrolled on study were treated on study
Groups:
- Post Auto Transplant Maintenance Therapy: only one arm of study : all patients treated on study with same maintenance therapy
Period: Overall Study
Arm/Group | Post Auto Transplant Maintenance Therapy
Started | 30
Completed | 16
Not Completed | 14
Not completed — Withdrawal by Subject | 3
Not completed — Lack of Efficacy | 8
Not completed — new secondary cancer | 1
Not completed — post surgery complications | 2

BASELINE CHARACTERISTICS:
Population: all patients enrolled were treated on study
Groups:
- Post Autologous Transplant Maintenance: one treatment arm all patients enrolled on study
Arm/Group | Post Autologous Transplant Maintenance
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30
number of participants treated [Count of Participants; unit: Participants] | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events, Graded According to CTCAE Version 4.0
Description: Adverse events Toxicity during the 24 months plus one month of post autologous transplant maintenance therapy
Time Frame: 2 years plus one month
Measure: Count of Participants; unit: Participants
Groups:
- Post Autologous Transplant Maintenance: one arm = all enrolled MM patients got post autologous transplant maintenance therapy
Arm/Group | Post Autologous Transplant Maintenance
Number analyzed (Participants) | 30
Participants | 30

2. Secondary Outcome: Overall Survival
Description: all MM patients who got post autologous transplant study therapy
Time Frame: Median 4.6 years from start of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Post Autologous Transplant Maintenance
Number analyzed (Participants) | 30
Participants | 21

3. Secondary Outcome: Disease Free Survival
Time Frame: Median of 4.6 years from start of study therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Post Autologous Transplant Maintenance
Number analyzed (Participants) | 30
Participants | 11

ADVERSE EVENTS:
Time Frame: Median 4.6 years from start of therapy
Arm/Group | Post Autologous Transplant Maintenance
All-Cause Mortality (participants affected / at risk) | 9/30
Serious Adverse Events (participants affected / at risk) | 4/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Post Autologous Transplant Maintenance (N=30)
pneumonia with sepsis (Infections and infestations) | 1 (1) — hospitalization
Pneumonia without sepsis (Infections and infestations) | 1 (1) — hospitalization
RSV Upper respiratory tract infection (Infections and infestations) | 1 (1) — hospitalization
palpitations (Cardiac disorders) | 1 (1) — hospitalization
OTHER ADVERSE EVENTS (reported when occurring in more than 3.3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Post Autologous Transplant Maintenance (N=30)
hyperglycemia (Investigations) | 2 — grade 2
hypoglycemia (Investigations) | 1 — grade 2
lymphocyte decreased (Investigations) | 11 — grade 2
lymphocyte decreased (Investigations) | 10 — grade 3
phosphorus decreased (Metabolism and nutrition disorders) | 5 — grade 2
upper respiratory tract infection (Infections and infestations) | 4 — grade 2
WBC decreased (Investigations) | 10 — grade 2
WBC decreased (Investigations) | 6 — grade 3
Platelet decreased (Investigations) | 7 — grade 2
Platelet decreased (Investigations) | 2 — grade 3
Platelet decreased (Investigations) | 1 — grade 4
ANC decreased (Investigations) | 9 — grade 2
ANC decreased (Investigations) | 7 — grade 3
ANC decreased (Investigations) | 2 — grade 4
fatigue (General disorders) | 2 — grade 3
cellulitis (Infections and infestations) | 3 — grade 2
vomiting (Gastrointestinal disorders) | 1 — grade 2
rash (Skin and subcutaneous tissue disorders) | 1 — grade 2
rash (Skin and subcutaneous tissue disorders) | 2 — grade 3
anemia (Blood and lymphatic system disorders) | 4 — grade 2
anemia (Blood and lymphatic system disorders) | 1 — grade 3
hypokalemia (Metabolism and nutrition disorders) | 1 — grade 2
Creatinine increased (Investigations) | 2 — grade 2
ALT increased (Investigations) | 1 — grade 2
diarrhea (Gastrointestinal disorders) | 1 — grade 2
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 — grade 2
albumin decreased (Metabolism and nutrition disorders) | 1 — grade 2
insomnia (Psychiatric disorders) | 1 — grade 2
Hypertension (Vascular disorders) | 1 — grade 2
hypertension (Vascular disorders) | 1 — grade 3
giardia gastrointestinal infection (Infections and infestations) | 1 — grade 2
superficial vein blood clot (Vascular disorders) | 1 — grade 2
bronchitis (Infections and infestations) | 2 — grade 2
thrush oral (Infections and infestations) | 1 — grade 2
Zoster (Infections and infestations) | 1 — grade 2
urinary tract infection (Infections and infestations) | 1 — grade 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/82/NCT02619682/Prot_SAP_000.pdf